CLINICAL TRIAL: NCT05460403
Title: Adjuvant Radiotherapy for Patients With Esophageal Squamous Cell Carcinoma After R0 Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zefen Xiao, Prof., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: K201427
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; postoperative radiotherapy; adjuvant radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery alone: patients without adjuvant radiotherapy after R0 resection.
- Adjuvant Radiotherapy: patients treated with adjuvant radiotherapy after R0 resection.
  Interventions: Radiation: Adjuvant Radiotherapy

INTERVENTIONS:
Radiation: Adjuvant Radiotherapy — Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks within 12 weeks after surgery in the absence of disease progression or unacceptable toxicity.
  Groups: Adjuvant Radiotherapy

SUMMARY:
This retrospective study is exploring the treatment effect and toxicity of adjuvant radiotherapy in patients diagnosed with esophageal squamous cell carcinoma after R0 resection.

DETAILED DESCRIPTION:
Surgery is one of the most important curative approaches for esophageal cancer. In real-world clinical practice, over 50% of the patients receiving surgical resection as primary management. For patients treated with surgical resection without adjuvant therapy, the probability of local-regional recurrence ranged from 23.0% to 56.5%, accounting for 55.6%-84.5% of the disease recurrence. Once encountering disease recurrence, the subsequent prognosis could be dismal. The median survival time after postoperative disease recurrence ranged from 3 to 8 months. Postoperative radiotherapy (PORT) was one of the potential topical treatment approaches prolonging local-regional recurrence time or moreover, attaining superior disease-free survival (DFS) or overall survival (OS) in selected patients. It is essential to identify patients potentially benefit from PORT. Besides, there were few studies evaluating the impact of postoperative radiation dose to survival outcomes in patients receiving PORT. Whether the PORT-related local-regional recurrence free survival (LRFS) enhancement could convert to OS or DFS improvement is still vague. The current study aimed at evaluating the value of PORT in patients diagnosed with esophageal squamous cell carcinoma after R0 resection.

ELIGIBILITY:
Inclusion Criteria:

* KPS≥70
* Pathologically diagnosis of esophageal cancer
* Complete resection (R0 resection)

Exclusion Criteria:

* Diagnosed with other malignancy within 5 years before surgery
* Encountered recurrence or port-site implantation receiving palliative-intended radiotherapy
* Diagnosed with adenosquamous carcinoma or basal cell-like carcinoma
* Treated with PORT with uncertain radiation dose
* Treated with PORT with radiation dose > 60Gy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with esophageal squamous cell carcinoma after R0 resection were enrolled from January 1993 and December 2012.
Sampling Method: Non-Probability Sample
Enrollment: 3591 (Estimated)
Dates: Start 2022-04-23 (Actual); Primary Completion 2023-07-02 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 5 years
  From the date of surgery to the date of death or the most recent follow-up.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | up to 5 years
  From the date of surgery to the date of any evidence of disease recurrence (recurrence in the tumor bed, anastomotic orifice, or in the regional lymph nodes, or metastasis in distant lymph nodes or distant organs), death or the most recent follow-up.
Local-regional recurrence-free survival (LRFS) | up to 5 years
  From the date of surgery to the date of recurrence in the tumor bed, anastomotic orifice, regional lymph nodes or the most recent follow-up.
Distant metastasis (DM) | up to 5 years
  From the date of surgery to the date of metastasis in distant lymph nodes, distant organs or the most recent follow-up.

OTHER OUTCOMES:
Adverse events | up to 5 years
  From the date of surgery to the date of death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zefen Xiao, MD, Principal Investigator — Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Science
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Science, Beijing, Chaoyang, China

REFERENCES:
- [Background] Rice TW, Chen LQ, Hofstetter WL, Smithers BM, Rusch VW, Wijnhoven BP, Chen KL, Davies AR, D'Journo XB, Kesler KA, Luketich JD, Ferguson MK, Rasanen JV, van Hillegersberg R, Fang W, Durand L, Cecconello I, Allum WH, Cerfolio RJ, Pera M, Griffin SM, Burger R, Liu JF, Allen MS, Law S, Watson TJ, Darling GE, Scott WJ, Duranceau A, Denlinger CE, Schipper PH, Lerut TE, Orringer MB, Ishwaran H, Apperson-Hansen C, DiPaola LM, Semple ME, Blackstone EH. Worldwide Esophageal Cancer Collaboration: pathologic staging data. Dis Esophagus. 2016 Oct;29(7):724-733. doi: 10.1111/dote.12520. PMID 27731547
- [Background] Rice TW, Ishwaran H, Hofstetter WL, Kelsen DP, Apperson-Hansen C, Blackstone EH; Worldwide Esophageal Cancer Collaboration Investigators. Recommendations for pathologic staging (pTNM) of cancer of the esophagus and esophagogastric junction for the 8th edition AJCC/UICC staging manuals. Dis Esophagus. 2016 Nov;29(8):897-905. doi: 10.1111/dote.12533. PMID 27905172
- [Background] Hsu PK, Chen HS, Huang CS, Liu CC, Hsieh CC, Hsu HS, Wu YC, Wu SC. Patterns of recurrence after oesophagectomy and postoperative chemoradiotherapy versus surgery alone for oesophageal squamous cell carcinoma. Br J Surg. 2017 Jan;104(1):90-97. doi: 10.1002/bjs.10334. Epub 2016 Nov 15. PMID 27859017
- [Background] Parry K, Visser E, van Rossum PS, Mohammad NH, Ruurda JP, van Hillegersberg R. Prognosis and Treatment After Diagnosis of Recurrent Esophageal Carcinoma Following Esophagectomy with Curative Intent. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S1292-300. doi: 10.1245/s10434-015-4840-5. Epub 2015 Sep 3. PMID 26334295
- [Background] Blom RL, Lagarde SM, van Oudenaarde K, Klinkenbijl JH, Hulshof MC, van Laarhoven HW, Bergman JJ, Busch OR, van Berge Henegouwen MI. Survival after recurrent esophageal carcinoma has not improved over the past 18 years. Ann Surg Oncol. 2013 Aug;20(8):2693-8. doi: 10.1245/s10434-013-2936-3. Epub 2013 Apr 3. PMID 23549882
- [Background] Xiao ZF, Yang ZY, Liang J, Miao YJ, Wang M, Yin WB, Gu XZ, Zhang DC, Zhang RG, Wang LJ. Value of radiotherapy after radical surgery for esophageal carcinoma: a report of 495 patients. Ann Thorac Surg. 2003 Feb;75(2):331-6. doi: 10.1016/s0003-4975(02)04401-6. PMID 12607634
- [Background] Deng W, Yang J, Ni W, Li C, Chang X, Han W, Zhou Z, Chen D, Feng Q, Liang J, Lv J, Wang X, Wang X, Deng L, Wang W, Bi N, Zhang T, Li Y, Gao S, Xue Q, Mao Y, Sun K, Liu X, Fang D, Wang D, Li J, Zhao J, Shao K, Li Z, Chen X, Han L, Wang L, He J, Xiao Z. Postoperative Radiotherapy in Pathological T2-3N0M0 Thoracic Esophageal Squamous Cell Carcinoma: Interim Report of a Prospective, Phase III, Randomized Controlled Study. Oncologist. 2020 Apr;25(4):e701-e708. doi: 10.1634/theoncologist.2019-0276. Epub 2020 Feb 21. PMID 32083766
- [Background] Ni W, Yu S, Xiao Z, Zhou Z, Chen D, Feng Q, Liang J, Lv J, Gao S, Mao Y, Xue Q, Sun K, Liu X, Fang D, Li J, Wang D, Zhao J, Gao Y. Postoperative Adjuvant Therapy Versus Surgery Alone for Stage IIB-III Esophageal Squamous Cell Carcinoma: A Phase III Randomized Controlled Trial. Oncologist. 2021 Dec;26(12):e2151-e2160. doi: 10.1002/onco.13914. Epub 2021 Aug 19. PMID 34309117
- See also: It is a national center for cancer research and treatment. It is one of the clinical trial bases approved by the Food and Drug Administration of State (SFDA) — http://www.cicams.ac.cn